CLINICAL TRIAL: NCT05780346
Title: Pilot Trial of Mentalizing-Focused Parenting Groups for Caregivers of Gender Diverse Youth
Brief Title: TGNB CARE Mentalizing-Focused Parenting Groups (TGNB-CARE)
Acronym: TGNB-CARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources and personnel available to complete study
Sponsor: Montefiore Medical Center (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14551
Record Dates: First submitted 2023-02-13; First posted 2023-03-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Parent-Child Relations
Keywords: Parenting; Gender Diverse; children

STUDY DESIGN:
Intervention Model Description: The proposed pilot study will include four treatment groups of 6 caregivers (N = 24) receiving the 12-session, 60-minute, video telehealth group intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARE Parenting Group Treatment (Experimental): Participants (i.e., caregivers of gender diverse youth) receive the CARE mentalizing-focused group parenting intervention.
  Interventions: Other: TGNB-CARE (Connecting and Reflecting Experience)

INTERVENTIONS:
Other: TGNB-CARE (Connecting and Reflecting Experience) — 12 session 60-minute mentalizing-focused parenting group with approximately 6 caregivers, facilitated by a mental health clinician

SUMMARY:
The primary objective of this pilot intervention study is to build upon the Connecting and Reflecting Experience (CARE) clinical trial [Clinical Trials Number: NCT04580459] and evaluate the acceptability, feasibility, and preliminary outcomes of CARE when implemented via tele-health among caregivers of transgender and nonbinary (TGNB) youth (TGNB-CARE).

The main questions it aims to answer are:

* To determine the feasibility and acceptability of the CARE treatment adaptation for caregivers of TGNB youth following the 12-session, mentalizing-focused, group parenting intervention. The study team hypothesizes that the adaptation and implementation of the CARE intervention will be found to be feasible and acceptable for study participants.
* To assess whether self-reported parenting stress and stressors, parental acceptance, parental reflective functioning, parent positive feelings, and perceived interpersonal support improve among study participants following the 12-session, mentalizing-focused, group parenting intervention. The study team hypothesizes that the CARE treatment group adaptation will show improvements across these outcomes.

Caregivers will be asked to complete surveys at baseline (T0), following their first session (T1), and at post-intervention (T2). A feedback interview will also be completed at T2.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers (mothers, fathers, primary caregivers, or legal guardians) who are English-speaking (as the research assessments and intervention will be conducted in English).
* Participants will be caregivers who:

  1. have a TGNB child who is receiving psychiatric services, has a mental health diagnosis, and/or has a diagnosis of gender dysphoria and is receiving medical or behavioral health services through Montefiore Medical Center and
  2. express interest in receiving a parenting intervention delivered via telehealth services through Montefiore Medical Center.

In addition, subjects will:

1. endorse past or current tension and/or interpersonal stress related to their child's gender identity and/or
2. express interest in receiving support in the context of gender-affirming parenting.

Exclusion Criteria:

* Caregiver has severe mental illness or significant cognitive impairment
* Additionally, caregivers who have participated in prior or current CARE groups or have participated in any parenting support groups in the past year will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Change in parenting stress | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parenting stress will be measured by administration of a caregiver self-report survey, the Parenting Stress Index, Fourth Edition, Short Form (PSI-4-SF). The PSI-4-SF is a 36-item survey divided into three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC), which combine to form a Total Stress scale. Items are rated on a 5-point Likert scale from "strongly disagree" (1) to "strongly agree" (5), then summed to yield subscale scores ranging from 12 to 60 and total scores ranging from 36 to 180. Raw scores can be converted to percentile based on a normed sample. Higher raw and percentile scores indicate higher levels of parenting stress. Scores falling between the 16th and 84th percentiles are considered within the normal range of parenting stress, scores between the 85th and 89th percentiles are considered high, and scores at the 90th percentile and above are considered in the clinically significant range.
Change in parental stressors | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parental stressors will be measured by administration of a caregiver self-report, The Stressors on Families of Trans Youth Checklist (SFTYC). Each item that is endorsed by the caregiver as having occurred is scored as '1' (excluding the 'none of the above' option on the form). If the caregiver endorses 'something else' on the form, each incident mentioned that is not already captured in existing checklist items is scored an additional '1'. The sum total of the endorsed items is the final score for this measure. Higher overall scores are indicative of higher external stressors on families/caregivers.
Change in parental acceptance of the gender-diverse child | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parental acceptance of the gender-diverse child will be assessed by administration of a caregiver self-report on the demographic questionnaire.
Change in parental reflective functioning | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parental reflective functioning as measured by parent/caregiver report on the Parental Reflective Functioning Questionnaire. Responses are reported on a 7-point Likert scale from 1 to 7. Total scores for the three sub-scales (Pre-Mentalizing Modes, Certainty about Mental States, and Interest and Curiosity) range from 6 to 42. Lower scores on Pre-Mentalizing Modes, moderate scores on Certainty about Mental States, and higher scores on Interest and Curiosity indicate better outcomes..
Change in Parental positive feelings about having a gender diverse child | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parental positive feelings about having a gender diverse child will be measured by administration of a caregiver self-report using the Trans Youth Can! Parent Positive Feelings Checklist (TYC-PPFC). Each item that is endorsed by the respondent as having occurred is scored as '1'. If the caregiver endorses 'something else', each incident mentioned that is not already captured in existing checklist items is scored an additional '1'. The sum total of the endorsed items is the final score for this measure. Higher overall scores are indicative of more positive feelings parents/caregivers of trans and non-binary youth experience in regard to their youth's gender.
Change in parental worries about having a gender diverse child | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in parental worries about having a gender diverse child will be measured by administration of a caregiver self-report using the Trans Youth Can! Parent Positive Feelings Checklist (TYC-PWC). Each item that is endorsed by the respondent as having occurred is scored as '1' (excluding the 'I have no great concerns' option which is coded as '0' and must be a unique choice if selected). If the caregiver endorses 'something else', each incident mentioned that is not already captured in existing checklist items is scored an additional '1'. The sum total of the endorsed items is the final score for this measure. Higher overall scores are associated with more potential factors that may concern parents/caregivers of trans and non-binary youth with regard to the youth's gender.
Change in perceived interpersonal support | Baseline (T0) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in perceived interpersonal support will be measured by administration of a caregiver self-report using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. All items are scored on a 7-point Likert scale, from 1 (Very Strongly disagree) to 7 (Very Strongly agree). Higher overall scores are associated with caregivers who perceive to receive greater interpersonal support from their social network.

OTHER OUTCOMES:
Intervention Feasibility | Following First CARE group session (T1) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Intervention feasibility will be measured by Feasibility of Intervention Measure (FIM). The FIM is a 4-item subscale that measures the extent to which a new treatment or innovation can be successfully used or carried out by the caregiver in this setting. All items are scored on a 5-point Likert scale, from 1 (Completely disagree) to 5 (Completely agree). Higher scores correlate with greater feasibility of the implementation of the intervention.
Intervention Acceptability | Following First CARE group session (T1) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Intervention acceptability will be measured by Acceptability of Intervention Measure (AIM). The AIM is a 4-item subscale that measures the extent to which a new treatment or innovation is found to be acceptable by the caregiver within this setting. All items are scored on a 5-point Likert scale, from 1 (Completely disagree) to 5 (Completely agree). Higher scores correlate with greater acceptability of the intervention.
Intervention Appropriateness | Following First CARE group session (T1) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Intervention appropriateness will be measured by Intervention Appropriateness Measure (IAM). The IAM is a 4-item subscale that measures the extent to which a new treatment or innovation is deemed to be appropriate by the caregiver within this setting. All items are scored on a 5-point Likert scale, from 1 (Completely disagree) to 5 (Completely agree). Higher scores correlate with greater appropriateness of the intervention.
Changes in therapeutic group cohesiveness | Following first CARE group session (T1) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Change in therapeutic group cohesiveness will be assessed using the self-reported Cohesiveness subscale of the Therapeutic Factors Inventory (TFI-COH). The Therapeutic Factors Inventory is a larger battery with 11 different subscales, developed to measure the therapeutic factors in group psychotherapy. The TFI-COH subscale used in the current study specifically assesses participant experiences of bondedness, acceptance, and mutual liking and trust within a particular therapy group. The TFI-COH includes nine items rated on a 7-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (7). Two items are reverse scored and then summed with remaining items to yield total scores ranging from 9 to 63. Higher total scores are generally indicative of perceptions of greater (more positive) cohesiveness within the therapy group.
Change in working alliance | Following First CARE group session (T1) and at post-intervention following completion of 12-session, 60-minute interventions (T2), an average of 18 weeks following session 1 of group
  Changes in therapeutic process variables will also be assessed using the using the Working Alliance Inventory - Short Form Revised (WAI-SR) scale. The WAI-SR is a 12-item patient-rated questionnaire that measures three domains of therapeutic alliance: agreement between patient and therapist on the goals of the treatment (Goal); agreement between patient and therapist about the tasks to achieve these goals (Task); and the quality of the bond between the patient and therapist (Bond). All items are scored on a 5-point Likert scale ranging from 1 ('rarely' or 'never') to 5 ('always'). Higher scores indicate a better therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda N Zayde, PsyD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No